CLINICAL TRIAL: NCT00236886
Title: Prospective Pilot Study on Metabolism and Weight Changes in Subjects With Diagnosed Partial Onset Epilepsy, With or Without Secondarily Generalized Seizures and Treated With Topiramate.
Brief Title: Prospective Pilot Study on Metabolism and Weight Changes in Topiramate-Treated Epilepsy Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR003703
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Epilepsy; Epilepsies, Partial; Epilepsy, Generalized; Seizures
Keywords: Epilepsy; Partial Epilepsy; Secondary Generalized Epilepsy; Primary Generalized Epilepsy; Tonic-Clonic Seizures; Topiramate; Weight Loss
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial; Epilepsy, Generalized; Seizures; Epilepsy, Idiopathic Generalized; Weight Loss | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to assess a possible predictor for weight loss seen in epilepsy patients treated with topiramate.

DETAILED DESCRIPTION:
Topiramate has been shown to be an effective anti-epileptic medication with a good safety profile. In clinical trials, some patients have experienced substantial weight loss. This prospective single center, open, pilot study will investigate whether there is any metabolic predictor for the weight loss. The patients will receive daily oral dose of topiramate in addition to anti-epileptic medications already prescribed by their physicians. A battery of metabolic tests including Body Mass Index (BMI), lean body mass, blood lipids and fasting glucose in tandem with other examinations will be taken before dispensing of topiramate, after 3 months and at the final visit. The study hypothesis is metabolic test results will provide a predictor of weight loss with topiramate. Patients will receive between 25 to 400mg daily of topiramate by mouth in addition to current anti-epileptic medications for up to 1 year. Dose will be adjusted (up to 1000 mg daily) by the investigators depending on the patients' clinical response.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of partial onset epilepsy, with or without secondary generalization. Patients with a diagnosis of epilepsy characterized by primary generalized tonic-clonic seizures may also qualify
* Currently taking one or more anti-epileptic medications on a stable dose for one month
* Weight between 40 and 130 kg (88 to 286 lbs)
* Female patients must be postmenopausal for at least 1 year, surgically incapable of childbearing, practicing an acceptable method of contraception (requires negative pregnancy test).

Exclusion Criteria:

* Patients with rapidly progressive disorders that may impair their weight or their reliable participation in the study
* Patients prone to severe malabsorption and/or metabolic disorders
* Patients who have mental retardation or impairment which would confound the interpretation of this study
* History (within the past six months) of a psychiatric or mood disorder requiring medical treatment
* History of poor compliance with past anti-epileptic drug therapy
* Suicide attempt in the past five years

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 1998-05; Study Completion 2000-06 (Actual)

PRIMARY OUTCOMES:
Metabolic test battery including Body Mass Index (BMI), lean body mass, blood lipids and fasting glucose along with physical examinations (including body weights) will be recorded at the beginning of the trial, after 3 months and after one year

SECONDARY OUTCOMES:
Safety evaluations (vital signs, physical exams, electrocardiogram, incidence and severity of adverse events) will be conducted throughout the study; Seizure frequency will be monitored throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Ben-Menachem E, Axelsen M, Johanson EH, Stagge A, Smith U. Predictors of weight loss in adults with topiramate-treated epilepsy. Obes Res. 2003 Apr;11(4):556-62. doi: 10.1038/oby.2003.78. PMID 12690085